CLINICAL TRIAL: NCT01808443
Title: Cryotherapy Versus Laser for the Treatment of Nongenital Cutaneous Warts: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Laser Versus Cryotherapy in the Treatment of Warts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The 306 Hospital of People's Liberation Army (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Shichao Lu, M.D., The 306 Hospital of People's Liberation Army
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 306PLA-001
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Warts
Keywords: cryotherapy; laser; cutaneous warts
MeSH Terms: conditions — Warts | interventions — Cryotherapy; Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryotherapy (Active Comparator): Cryotherapy, at most 4 times
  Interventions: Other: Cryotherapy
- laser (Experimental): laser, at most 4 times
  Interventions: Other: laser

INTERVENTIONS:
Other: Cryotherapy — up to a maximum of four treatments every 21-28 days
  Arms: Cryotherapy
Other: laser — up to a maximum of four treatments every 21-28 days
  Arms: laser

SUMMARY:
The purpose of this study is to test the efficacy of laser versus cryotherapy on the treatment of warts

DETAILED DESCRIPTION:
Cutaneous warts were a common skin diseases caused by human papilloma virus (HPV) infection. Although warts may spontaneously resolve, many patients seek for treatment for various reasons. There are many kinds of treatments for cutaneous warts, including salicylic acid, cryotherapy, laser, etc. A recent high quality RCT confirmed that the cure rate of topical salicylic acid and frozen has no difference at six months, but the efficacy of laser versus cryotherapy on the treatment of warts remains unclear. Therefore, we designed a randomized controlled trial to test the efficacy of laser versus cryotherapy on the treatment of warts.

ELIGIBILITY:
Inclusion Criteria:

* Patients have cutaneous warts, including common warts(d≥1cm or n≥5 ), plantar warts, periungual warts, mosaic warts, which are suitable for cryotherapy and laser treatment .
* patients aged eighting years and over, who have junior school degree or above

Exclusion Criteria:

* Patients who have more than 20 warts
* Patients who are currently participating in another trial for the treatment of their warts
* Patients who took immunosuppressant drugs such as oral corticosteroids within the past three months.
* Patients who are pregnant or ready for pregnancies or breast-feeding.
* Patients who have impaired healing eg due to diabetes, vascular disease, vitamin A deficiency, hyperthyroidism and hypothyroidism.
* Patients who have autoimmune diseases, eg SLE, dermatomyositis, scleroderma and other diseases .
* Patients who have cold intolerance, eg cold urticaria, cryoglobulinaemia, cold agglutinin syndrome, Raynaud's syndrome.
* Patients who have local injections intolerance.
* Patients who have local hypoesthesia .
* Patients who can not tolerate cryotherapy or laser treatment for their own reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
cure rate | Cure rate will be calculated at 16 weeks and 6 months from the first treatment
  Warts was considered cured if they was no longer visible and could not be palpated anymore by hand. Assessment of whether or not cured was performed on site by a senior dermatologist

SECONDARY OUTCOMES:
effective rate | Effective rate will be calculated at 16 weeks from the first treatment
  Effective assessment is performed by a senior dermatologist.
recurrence rate | Recurrence rate will be calculated at 12 months from the first treatment
  A wart was considered recurrence if there are abnormalities or palpated foreign body in the original place.
average cure days | Average cure days will be calculated at 6 months from the first treatment
  Cure days was defined as the period from the first treatment until the date of clearance.
side effects | Side effects will be assessed within 3-4 weeks after each treatment
  including pain, swelling, blisters, blood blisters, bruising, bleeding,scarring, hypopigmentation, hyperpigmentation.
pain intensity | Pain intensity will be assessed within 3-4 weeks after each treatment
  on a scale of 0-10, where 0 is no pain and 10 is extremely painful
patient satisfaction | Patient satisfactionwill be assessed within 3-4 weeks after each treatment
  on a five-point scale, from 'very satisfied' to 'very satisfied'
treatment costs | Treatment costs will be recorded within 10 minutes after each treatment
  record the cost after each treatment
relationship between HPV type and curative effect | Relationship between HPV type and curative effect will be analyzed at 16 weeks and 6 months from the first treatment
  take a small amount of cutaneous warts lesions and extract HPV DNA before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shichao Lu, MD, Principal Investigator — Dermatology Deparment of the 306 Hospital of PLA
Locations (1):
- The 306 Hospital of PLA, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided